CLINICAL TRIAL: NCT02334280
Title: Evaluation of A Statewide Program to Prevent Early Mortality and to Promote Fitness in Persons With SMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: InSHAPE Implementation Study
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder
Keywords: Community mental health; Health coach; Weight loss; Fitness; Serious mental illness; Health promotion
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In SHAPE (Experimental): In SHAPE is a health promotion intervention consisting of a fitness club membership and a health promotion coach with basic certification as a fitness trainer, instruction on principles of healthy eating and nutrition, and training in tailoring individual wellness plans to the needs of persons with serious mental illness.
  Interventions: Behavioral: In SHAPE
- Usual-Care Control (No Intervention): Usual-care consumers agreed to delay participation in In SHAPE for 12 months.

INTERVENTIONS:
Behavioral: In SHAPE — In SHAPE is a health promotion intervention consisting of a fitness club membership and a health promotion coach with basic certification as a fitness trainer, instruction on principles of healthy eating and nutrition, and training in tailoring individual wellness plans to the needs of persons with serious mental illness.
  Arms: In SHAPE

SUMMARY:
The goal of this project, which has not changed, is to evaluate the statewide implementation of a two-component intervention (health promotion plus academic detailing) with respect to consumer outcomes and changes in provider prescribing. The intervention, called In SHAPE, is delivered to people with serious mental illness (SMI) by two community mental health clinics (CMHCs). These CMHCs are compared to two CMHCs delivering usual-care to individuals with SMI. The specific aims of this study are:

1. Evaluate person-level and provider-level outcomes including: (a) consumer health behaviors, health indicators, mental health indicators, and acute health service utilization, (b) provider prescribing practices and program fidelity, and (c) program costs.
2. Evaluate system-level outcomes including: (a) consumer health behaviors and health indicators, (b) provider prescribing and program fidelity, and (c) acute services use.

DETAILED DESCRIPTION:
Individuals with SMI die 10-25 years earlier than the general population and have disproportionately greater rates of medical comorbidity and disability associated with high rates of obesity, sedentary lifestyle, metabolic syndrome, and poor dietary habits. Despite greater costs and adverse outcomes associated with the combination of mental illness and poor physical health, little attention has been paid to the development of health promotion interventions designed to address the needs of the high-risk group of people with SMI. This natural experiment presents an unprecedented opportunity to evaluate the public health impact of a statewide health-promotion program for persons with SMI, a potential model for reducing early mortality among persons with SMI served by state mental-health systems nationwide.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Serious mental illness defined by (a) an axis I diagnosis of major depression, bipolar disorder, schizoaffective disorder, or schizophrenia, (b) moderate impairment across multiple areas of psychological functioning, or (c) Global Assessment of Functioning (GAF) score less than 61
* Able to provide voluntary informed consent for participation in the study by the participant or by the participant's legally designated guardian or conservator
* Poor fitness as indicated by BMI > 25 or failure to adhere to the US Department of Health and Human Services Physical Activity Guidelines for Americans, i.e., at least 2.5 hr/week of moderate or 75 min/week of vigorous activity in more than one session
* Medical clearance for participation in an exercise and dietary modification program by a physician, physician assistant, or nurse practitioner
* An expressed willingness to participate in a diet and exercise program
* Currently taking an atypical antipsychotic medication
* Able to walk a city block
* Responsible for choice of foods and how they are prepared

Exclusion Criteria:

* Currently residing in a nursing home or group home
* Terminal physical illness expected to result in the death of the study subject within one year
* Primary diagnosis of dementia, co-morbid diagnosis of dementia, or significant cognitive impairment as indicated by a Mini-Mental State Examination (MMSE) score < 24
* Inability to speak and understand English
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in exercise capacity | baseline, 6-, 12-, and 24-months
  Change in exercise capacity measured by the 6-minute walk test.

SECONDARY OUTCOMES:
Self-reported physical activity | baseline, 6-, 12-, and 24-months
  Change in self-reported physical activity measured with International Physical Activity Questionnaire (IPAQ)
Change in dietary behaviors | baseline, 6-, 12-, and 24-months
  Change in dietary behaviors measured with the Block Food Frequency Questionnaire (FFQ)21 and the Questionnaire on Eating and Weight Patterns (QEWP).
Change in stage of change | baseline, 6-, 12-, and 24-months
  Change in stage of change measured with the Weight Loss Behavior-Stage of Change Scale (WLB-SOC) 23 to assess stage of change for engaging in healthy eating and exercise behaviors.
Change in eating behavior | baseline, 6-, 12-, and 24-months
  Change in eating behavior measured with the Dutch Eating Behavior Questionnaire which includes 13 questions assessing emotional eating and 10 questions related to external eating behaviors
Change in physical measurement | baseline, 6-, 12-, and 24-months
  Including height, weight, pulse, CO2 level, lung capacity from spirometer, variables from impedance measure such as percentage of body fat and percentage of lean muscle mass, cholesterol and triglyceride levels from finger stick (cholesterol data for data points that have already passed will be collected from participants' clinic and hospital records), waist circumference: BMI derived from height and weight.
Change in smoking and substance use | baseline, 6-, 12-, and 24-months
  Change in smoking and substance use measured by questions developed for R01DA021245, "Smoking Cessation and Smoking Relapse Prevention in Patients with Schizophrenia," and questions from the "Quit Smoking Decision Aid"( developed by Ferron and Brunette, CPHS # 180) to ascertain smoking frequency, quantity, and cessation attempts
Change in psychological functioning (depression, negative symptoms, and self-efficacy). | baseline, 6-, 12-, and 24-months
  Change in psychological functioning measured by the Center for Epidemiologic Studies Depression Scale,Scale to Assess Negative Symptoms,16 and the Self-Rated Abilities for Health Practices Scale will be used to assess these constructs.
Change in social functioning | baseline, 6-, 12-, and 24-months
  Change in social functioning measured by the Social Network Questionnaire and Lehman Social Contact Scale.
Change in family contact | baseline, 6-, 12-, and 24-months
  Change in family contact measured by the Revised Family Contact Questionnaire.
Change in social support and eating habits | baseline, 6-, 12-, and 24-months
  Change in the impact of social support on eating habits measured by the Social Support and Eating Habits Survey
Change in social support and exercise | baseline, 6-, 12-, and 24-months
  Change in the impact of social support on exercise behaviors measured by the Social Support and Exercise Survey
Change in comorbid medical illness | baseline, 6-, 12-, and 24-months
  Change in comorbid medical illness measured using a medical problems list.
Change in medications | baseline, 6-, 12-, and 24-months
  Change in medications measured by gathering information from participants about type, dose, and frequency of all prescribed medications.
Change in service use | baseline, 6-, 12-, and 24-months
  Measured change in service use based on a measured designed for the In SHAPE studies to collect self-reported use of emergency services and hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bartels, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - West Central Behavioral Health, Lebanon, New Hampshire
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Greater Nashua Mental Health Center at Community Council, Nashua, New Hampshire
  - Center for Life Management, Salem, New Hampshire